CLINICAL TRIAL: NCT00372138
Title: Prevention of Endoleaks Using Autologous Platelet Gel During Endovascular Procedures on Unruptured Abdominal Aortic Aneurysms: Pilot Study
Brief Title: Prevention of Endoleaks Using Autologous Platelet Gel on Unruptured Abdominal Aortic Aneurysms
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AFSSAPS TC211; LOC/05-04 (Other: Rennes University Hospital); CIC0203/057
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Abdominal Aortic Aneurysms
Keywords: Abdominal aortic aneurysms; Endoleaks; Prevention
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

ARMS (1):
- PRP + autologous thrombin (Experimental): simultaneous perioperative PRP and autologous thrombin in the aneurysm sac, during the endovascular treatment of unruptured abdominal aortic aneurysms
  Interventions: Procedure: PRP + autologous thrombin

INTERVENTIONS:
Procedure: PRP + autologous thrombin — simultaneous perioperative PRP and autologous thrombin in the aneurysm sac, during the endovascular treatment of unruptured abdominal aortic aneurysms

SUMMARY:
The main risk of aortic aneurysms is rupture that leads to a high risk of death. A preventive surgical treatment is thus needed. In order to reduce the morbidity and mortality associated with conventional surgery, an endovascular approach (insertion of an endovascular stent graft)is now widely favored. The main problem of this procedure is the occurrence of endoleaks (persistence of a communication between the aneurysm and the aorta). A new approach is proposed to prevent these endoleaks. The principle is to draw blood from the patient, separate the blood from the platelets, and reinject both platelet rich plasma (PRP) and autologous thrombin, in order to form a platelet gel (PRP + autologous thrombin). Before studying the efficacy of this technique, its safety of use and feasibility must be evaluated.

DETAILED DESCRIPTION:
The main risk of aortic aneurysms is rupture. Onset is usually sudden, leading to the death of the patient in 80% to 90% of cases. The elective treatment of abdominal aortic aneurysms, therefore, seems to be a priority. In order to reduce the morbidity and mortality associated with conventional surgery, an endovascular approach (insertion of an endovascular stent graft using the endovascular aneurysm repair procedure) is now widely favored. The main problem, during follow-up of patients wearing an endovascular stent graft, is the occurrence of endoleaks resulting in retrograde filling of the aneurysm sac. The ideal is to prevent these endoleaks either by new developments in endovascular stent grafts or by using adjuvant therapy during the procedure. The principle is to draw blood from the patient, separate the blood from the platelets, and reinject it into two separate catheters, one with platelet rich plasma (PRP) and the other with autologous thrombin, in order to form a platelet gel (PRP + autologous thrombin). Before studying the efficacy of this technique, its safety of use and feasibility must be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Patient eligible to endovascular treatment:

* Any patient having an infrarenal or aortoiliac abdominal aortic aneurysm needing surgical treatment,
* With an infrarenal neck larger than 10 mm,
* No thrombi in the neck,
* Calcifications of the neck smaller than 30% of the circumference.
* The maximum diameter of the aneurysm must be at least 50 mm and/or an annual growth rate of more than 10 mm and/or if the aneurysm is symptomatic,
* With no major tortuosity of the two iliac axes with an aortoiliac angle greater than 80°,
* An external iliac diameter of at least 8 mm,
* An angle between the interrenal aorta and the neck of 0-45°.
* The patient must meet at least one of the operability criteria of the French Health Products Safety Agency (AFSSAPS)

Exclusion Criteria:

* Patient with a hemostatic disorder, previously known or discovered during the preoperative lab work-up,
* Patient whose arterial anatomy is incompatible with the criteria form use of a TALENT type endovascular stent graft,
* Patient with an aneurysm whose rapid progression (risk of rupture) does not allow a radiological and scanographic assessments to be performed,
* Patient allergic to the iodized contrast media,
* Disease of the connective tissue (Marfan's Syndrome) or inflammatory aneurysm,
* Patient with an aneurysm that includes the orifice of both internal iliacs,
* Patient in whom it is essential to keep the inferior mesenteric artery permeable,
* Patient surgically converted after failure of an endovascular technique,
* Pregnant women,
* Failure of stent graft insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2007-10 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety of the perioperative procedure for injecting PRP + autologous thrombin assessed by distal embolism, colic necrosis, aneurysm rupture. | perioperative
  * systemic hemodynamics (systolic, diastolic, and mean arterial pressure, before and after insertion of the endovascular stent graft, after insertion of the 2 injection catheters, and 1, 5, and 15 minutes after injection of the thrombin and PRP),
  * pressure inside the aneurysm 5 minutes after injection with the thrombin and PRP,
  * endoleaks at end of surgery,
  * distal embolism, colic necrosis,
  * rupture of the aneurysm,
  * prosthetic migration
  * plication, stenosis of the stent graft
  * thrombosis of the stent graft,
  * occlusive arterial lesion

SECONDARY OUTCOMES:
Description of the perioperative surgical technique for injecting PRP + autologous thrombin | perioperative
  * length of the procedure,
  * insertion of the two injection catheters,
  * preparation of the platelet gel,
  * problem encountered during injection of the gel
Rate of occurrence of endoleaks at 1 month and types of endoleaks, | 1 month
Time to onset of endoleaks, | 1 month
Rate of complications related to the endovascular procedure. | 1 month
- Rate of early postoperative complications (< 30 days) | < 30 days
  * distal embolism, colic necrosis,
  * rupture of the aneurysm,
  * prosthetic migration,
  * plication, stenosis of the stent graft,
  * thrombosis of the stent graft,
  * occlusive arterial lesion,
  * reoperation and reason for reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Alain Cardon, MD, Principal Investigator — CHU Rennes; Bruno Laviolle, MD, Study Chair — CHU Rennes
Locations (1):
- Service de Chirurgie Vasculaire - Hôpital de Pontchaillou, Rennes, France